CLINICAL TRIAL: NCT00357019
Title: Study of the Clinical and Biological Efficacity of NAAXIA SINE® in Vernal Keratoconjunctivitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laboratoires Thea (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TPO 09/99 NAAXIA SINE Phase IV
Record Dates: First submitted 2006-07-26; First posted 2006-07-27 (Estimated); Last update posted 2006-07-27 (Estimated); Status verified 2006-07

CONDITIONS: Keratoconjunctivitis, Vernal
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — isospaglumic acid

INTERVENTIONS:
Drug: N-acetyl-aspartyl-glutamate (NAAXIA Sine)

SUMMARY:
To assess the clinical and biological efficacity of preservative free NAAGA eyes drops in vernal keratoconjunctivitis

DETAILED DESCRIPTION:
The objective of this pilot study is to evaluate the clinical and biological efficacy of preservative free NAAGA eyedrops in VKC -by in particular the levels of ECP and MPO in tears- comparatively to the activity of levocabastine eyedrops.

ELIGIBILITY:
Inclusion Criteria:

* Patients with vernal keratoconjunctivitis,
* mild or moderate : clinical score >3 and <= 14, calculated from 4 major symptoms (itching, tearing, photophobia, foreign body sensation) and 6 major clinical signs (conjunctival erythema, conjunctival chemosis, discharge, papillae, limbal infiltrates and corneal epithelial disease)
* age >= 4 years old

Exclusion Criteria:

* no occurrence of ocular trauma or infection (within the 3 months preceding the study),
* no ocular medical treatment (topical or not) within the 5 days preceding the study,
* no ocular laser (within the 3 previous months),
* no ocular surgery (within the previous year),
* patient who signs the informed consent form (or his/her parents or legal guardian in the case of underage patient).

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-04; Study Completion 2002-10

PRIMARY OUTCOMES:
ECP tear concentration

SECONDARY OUTCOMES:
Tolerance

CONTACTS AND LOCATIONS:
Overall Officials: Andréa LEONARDI, Professor, Principal Investigator — Clinica Oculistica, Padova (Italy)

REFERENCES:
- [Derived] Leonardi A, Bremond-Gignac D, Bortolotti M, Violato D, Pouliquen P, Delval L, Grouin JM, Fregona IA. Clinical and biological efficacy of preservative-free NAAGA eye-drops versus levocabastine eye-drops in vernal keratoconjunctivitis patients. Br J Ophthalmol. 2007 Dec;91(12):1662-6. doi: 10.1136/bjo.2007.117515. Epub 2007 Jun 21. PMID 17585003